CLINICAL TRIAL: NCT00697190
Title: Clinical Performance of Atypical Contact Lens Powers on Subjects With Astigmatism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR-4523
Record Dates: First submitted 2008-06-10; First posted 2008-06-13 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- senofilcon A/galyfilcon A (Active Comparator): senofilcon A silicone hydrogel toric contact lenses will be worn first. galyfilcon A silicone hydrogel toric contact lenses will be worn second.
  Interventions: Device: senofilcon A toric; Device: galyfilcon A toric
- galyfilcon A/senofilcon A (Active Comparator): galyfilcon A silicone hydrogel toric contact lenses worn first. senofilcon A silicone hydrogel toric contact lenses worn second.
  Interventions: Device: senofilcon A toric; Device: galyfilcon A toric

INTERVENTIONS:
Device: senofilcon A toric — silicone hydrogel contact lens for patients with astigmatism
  Other Names: Acuvue Oasys for Astigmatism
Device: galyfilcon A toric — silicone hydrogel contact lens for patients with astigmatism
  Other Names: Acuvue Advance for Astigmatism

SUMMARY:
This study will evaluate the fitting characteristics and physiological response of two toric lenses manufactured by Vistakon.

ELIGIBILITY:
Inclusion Criteria:

* Able to wear study lenses in parameters available.
* At least 18
* understand and sign informed consent
* willing to follow the protocol
* achieve at least 6/9 Visual Acuity (VA), both eyes (OU) with study lenses
* hyperopes: +2.00 to +4.00 with -0.75 D cylinder around 180, high myopes: -6.00 to -8.00 with -1.25 D cylinder around 180
* oblique axis: -2.00 to -4.00 with -0.75 D cyl around 45 or 135, have worn Soft Contact Lenses's within last 6 months

Exclusion Criteria:

* Any ocular or systemic disorder which may contraindicate Contact Lens (CL) wear
* any topical ocular medication
* aphakic
* corneal refractive surgery,
* corneal distortion from hard CL wear or keratoconus
* pregnant or lactating
* grade 2 or worse slit lamp signs
* infectious disease
* previous clinical study within 2 weeks
* don't agree to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Eurolens Research, Manchester, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: First Intervention
Arm/Group | Senofilcon A/Galyfilcon A | Galyfilcon A/Senofilcon A
Started | 19 | 20
Completed | 19 | 20
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Senofilcon A/Galyfilcon A | Galyfilcon A/Senofilcon A
Started | 18 (one subject moved away between the first period and second period.) | 20
Completed | 18 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Completed Subjects: All subjects that completed the study were analyzed. One subject from the senofilcon A/ galyfilcon A arm dropped from the study between the first and second intervention. The subject moved out of town.
Arm/Group | All Completed Subjects
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 11
Region of Enrollment [Number; unit: participants]
  United Kingdom | 38

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Conjunctival Hyperemia in Subjects That Are High Myopes (Have a High Degree of Nearsightedness)
Description: Conjunctival hyperemia measures the redness across the white of the eye. The investigator used a grading scale of 0=none, 1=slight, 2=moderate, 3=severe.
Time Frame: after 6 hours of wear
Population: There were 11 subjects that were high myopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Senofilcon A: This group represents all high myope subjects that completed the study and wore senofilcon A toric contact lenses as first or second intervention.
- Galyfilcon A: This group represents all high myope subjects that completed the study and wore galyfilcon A toric contact lenses as first or second intervention.
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 11 | 11
Units on a scale | 1.10 (0.05) | 1.23 (0.05)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senoflicon A toric is non-inferior to galyfilcon A toric in conjunctival hyperemia; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.13, 97.5% CI 2-sided [-0.29 to 0.04], Standard Error of Mean 0.09 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

2. Primary Outcome: Assessment of Conjunctival Hyperemia in Subjects That Are Hyperopes (Farsighted)
Description: as for outcome 1
Time Frame: after 6 hours of wear
Population: There were 14 subjects that were hyperopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Senofilcon A: This group represents all hyperope subjects that completed the study and wore senofilcon A toric contact lenses as first or second intervention.
- Galyfilcon A: This group represents all hyperope subjects that completed the study and wore galyfilcon A toric contact lenses as first or second intervention.
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 14 | 14
Units on a scale | 1.16 (0.07) | 1.18 (0.05)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in conjunctival hyperemia; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.02, 97.5% CI 2-sided [-0.10 to 0.06], Standard Error of Mean 0.04 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

3. Primary Outcome: Assessment of Conjunctival Hyperemia in Subjects That Are Oblique Astigmats (Have an Abnormally Curved Cornea)
Description: as for outcome 1
Time Frame: after 6 hours of wear
Population: There were 13 subjects that were oblique astigmats within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Senofilcon A: This group represents all oblique astigmat subjects that completed the study and wore senofilcon A toric contact lenses as first or second intervention.
- Galyfilcon A: This group represents all oblique astigmat subjects that completed the study and wore galyfilcon A toric contact lenses as first or second intervention.
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 13 | 13
Units on a scale | 1.08 (0.07) | 1.14 (0.08)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in conjunctival hyperemia; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.07, 97.5% CI 2-sided [-0.23 to 0.10], Standard Error of Mean 0.08 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

4. Primary Outcome: Assessment of Limbal Hyperemia in Subjects That Are High Myopes (Have a High Degree of Nearsightedness)
Description: Limbal hyperemia measures the redness around the edge of the cornea. The investigator used a grading scale of 0=none, 1=slight, 2=moderate, 3=severe.
Time Frame: after 6 hours of wear
Population: There were 11 subjects that were high myopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 11 | 11
Units on a scale | 0.97 (0.05) | 1.07 (0.07)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in limbal hyperemia; Test type: Non-Inferiority or Equivalence — Non-inferior margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.11, 97.5% CI 2-sided [-0.25 to 0.04], Standard Error of Mean 0.08 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

5. Primary Outcome: Assessment of Limbal Hyperemia in Subjects That Are Hyperopes (Farsighted)
Description: as for outcome 4
Time Frame: after 6 hours of wear
Population: There were 14 subjects that were hyperopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 14 | 14
Units on a scale | 0.95 (0.06) | 1.00 (0.06)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in limbal hyperemia; Test type: Non-Inferiority or Equivalence — Non-inferior margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 97.5% CI 2-sided [-0.16 to 0.07], Standard Error of Mean 0.06 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

6. Primary Outcome: Assessment of Limbal Hyperemia in Subjects That Are Oblique Astigmats (Have an Abnormally Curved Cornea)
Description: as for outcome 4
Time Frame: after 6 hours of wear
Population: There were 13 subjects that were oblique astigmats within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 13 | 13
Units on a scale | 1.01 (0.08) | 1.06 (0.07)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in limbal hyperemia; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.06, 97.5% CI 2-sided [-0.25 to 0.14], Standard Error of Mean 0.10 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

7. Primary Outcome: Assessment of Corneal Staining in Subjects That Are High Myopes (Have a High Degree of Nearsightedness)
Description: Corneal staining measures changes to the surface of the cornea, as evaluated by the degree of staining with sodium fluorescein solution. The investigator used a grading scale of 0=none, 1=slight, 2=moderate, 3=severe.
Time Frame: after 6 hours of wear
Population: There were 11 subjects that were high myopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 11 | 11
Units on a scale | 0.40 (0.07) | 0.22 (0.05)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in corneal staining; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = 0.18, 97.5% CI 2-sided [0.04 to 0.32], Standard Error of Mean 0.07 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

8. Primary Outcome: Assessment of Corneal Staining in Subjects That Are Hyperopes (Farsighted)
Description: as for outcome 7
Time Frame: after 6 hours of wear
Population: There were 14 subjects that were hyperopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 14 | 14
Units on a scale | 0.19 (0.07) | 0.28 (0.09)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in corneal staining; Test type: Non-Inferiority or Equivalence — Non-inferior margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 97.5% CI 2-sided [-0.26 to 0.08], Standard Error of Mean 0.08 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

9. Primary Outcome: Assessment of Corneal Staining in Subjects That Are Oblique Astigmats (Have an Abnormally Curved Cornea)
Description: as for outcome 7
Time Frame: after 6 hours of wear
Population: There were 13 subjects that were oblique astigmats within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 13 | 13
Units on a scale | 0.35 (0.08) | 0.18 (0.08)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in corneal staining; Test type: Non-Inferiority or Equivalence — Non-inferior margin = 0.33; Mixed Models Analysis; Median Difference (Final Values) = 0.17, 97.5% CI [0.02 to 0.33], Standard Error of Mean 0.08 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

10. Primary Outcome: Assessment of Conjunctival Staining in Subjects That Are High Myopes (Have a High Degree of Nearsightedness)
Description: Conjunctival staining measures the changes to the conjunctival surface as evaluated by the degree of staining with sodium fluorescein solution. The investigator used a grading scale of 0=none, 1=slight, 2=moderate, 3=severe.
Time Frame: after 6 hours of wear
Population: There were 11 subjects that were high myopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 11 | 11
Units on a scale | 1.68 (0.09) | 1.69 (0.14)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in conjunctival staining; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.01, 97.5% CI 2-sided [-0.27 to 0.26], Standard Error of Mean 0.13 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

11. Primary Outcome: Assessment of Conjunctival Staining in Subjects That Are Hyperopes (Farsighted)
Description: as for outcome 10
Time Frame: after 6 hours of wear
Population: There were 14 subjects that were hyperopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 14 | 14
Units on a scale | 0.96 (0.10) | 1.17 (0.08)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in conjunctival staining; Test type: Non-Inferiority or Equivalence — Non-inferior margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.21, 97.5% CI 2-sided [-0.34 to -0.08], Standard Error of Mean 0.07 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

12. Primary Outcome: Assessment of Conjunctival Staining in Subjects That Are Oblique Astigmats (Have an Abnormally Curved Cornea)
Description: as for outcome 10
Time Frame: after 6 hours of wear
Population: There were 13 subjects that were oblique astigmats within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 13 | 13
Units on a scale | 1.12 (0.09) | 1.42 (0.08)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in conjunctival staining; Test type: Non-Inferiority or Equivalence — Non-inferior margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.34, 97.5% CI 2-sided [-0.54 to -0.15], Standard Error of Mean 0.10 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

13. Primary Outcome: Assessment of Papillary Conjunctivitis in Subjects That Are High Myopes (Have a High Degree of Nearsightedness)
Description: Papillary conjunctivitis measures the changes to the conjunctival surface on the underside of the upper eyelid. The investigator used a grading scale of 0=none, 1=slight, 2=moderate, 3=severe.
Time Frame: after 6 hours of wear
Population: There were 11 subjects that were high myopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 11 | 11
Units on a scale | 1.09 (0.07) | 1.08 (0.07)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in papillary conjunctivitis; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 97.5% CI 2-sided [-0.12 to 0.14], Standard Error of Mean 0.07 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

14. Primary Outcome: Assessment of Papillary Conjunctivitis in Subjects That Are Hyperopes (Farsighted)
Description: as for outcome 13
Time Frame: after 6 hours of wear
Population: There were 14 subjects that were hyperopes within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 14 | 14
Units on a scale | 1.12 (0.06) | 1.21 (0.09)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in papillary conjunctivitis; Test type: Non-Inferiority or Equivalence — Non-inferior margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 97.5% CI 2-sided [-0.23 to 0.05], Standard Error of Mean 0.07 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

15. Primary Outcome: Assessment of Papillary Conjunctivitis in Subjects That Are Oblique Astigmats (Have an Abnormally Curved Cornea)
Description: as for outcome 13
Time Frame: after 6 hours of wear
Population: There were 13 subjects that were oblique astigmats within the total completed population of 38.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Senofilcon A | Galyfilcon A
Number analyzed (Participants) | 13 | 13
Units on a scale | 1.01 (0.05) | 1.10 (0.04)
Statistical Analysis 1: Comparison: Senofilcon A vs Galyfilcon A; Alternative hypothesis is that senofilcon A toric is non-inferior to galyfilcon A toric in papillary conjunctivitis; Test type: Non-Inferiority or Equivalence — Non-inferior margin = 0.33; Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 97.5% CI 2-sided [-0.20 to 0.02], Standard Error of Mean 0.06 — The mean difference is calculated as senofilcon A toric minus galyfilcon A toric

ADVERSE EVENTS:
Groups:
- Senofilcon A: senofilcon A silicone hydrogel toric contact lenses worn in the first or second intervention.
- Galyfilcon A: galyfilcon A silicone hydrogel toric contact lenses worn in the first or second intervention.
Arm/Group | Senofilcon A | Galyfilcon A
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 1/19 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Senofilcon A (N=19) | Galyfilcon A (N=20)
asymptomatic infiltrative event (Eye disorders) | 1 (1) | 0 (0)
non-significant corneal infiltrate event (Eye disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may not publish, divulge, reveal, disclose, or use the data and or results of the study without prior written consent of Vistakon.